CLINICAL TRIAL: NCT05853224
Title: An Interventional, Pre-Market, Double-Blinded, Controlled, Two Stages Study to Evaluate the Safety and Performance of Crosslinked Hyaluronic Acid Hydrogel (With and Without Lidocaine) for the Treatment of Soft Tissue Deficits
Brief Title: An Interventional Study to Evaluate the Safety and Performance of Crosslinked Hyaluronic Acid Hydrogel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biopolimeri Srl (Industry)
Collaborators: 1Med (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS-14-01
Record Dates: First submitted 2023-03-28; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Dermal Filler; Volume Deficiency of the Midface
Keywords: Volume Loss, Aging, Aesthetic

STUDY DESIGN:
Intervention Model Description: Each Subject, after signing the Informed Consent (ICF), will enter into a screening phase during which the baseline tests will be conducted.
  At baseline visit (V0), according to the Instruction For Use (IFU) and to Investigator's judgment based on the patient's starting clinical situation, the subject will be treated with one of the three variants of Crosslinked Hyaluronic Acid (CLHA) Hydrogel as indicated below:
  * CLHA Hydrogel 26 mg/ml (with and without lidocaine) will be injected in the hypodermis of the nasolabial folds (NLFs);
  * CLHA Hydrogel 20 mg/ml (with and without lidocaine) will be injected in the lips mucosa/submucosa;
  * CLHA Hydrogel 18 mg/ml (with and without lidocaine) will be injected in the superficial dermis of the perioral lines.
Who Masked: Participant, Outcomes Assessor
Masking Description: The study will be double-blinded: patients and the treating investigator will not know which variant of each product (with and without lidocaine) will be injected in the left/right side of the face (or in the upper/lower lip for CLHA Hydrogel 20 mg/ml) and the evaluating investigator will be different from the treating investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Crosslinked Hyaluronic Acid (CLHA) Hydrogel with Lidocaine (Experimental): Patients were treated, on one side of the face with crosslinked Hyaluronic Acid Hydrogel with 0.3% lidocaine hydrochloride.
  Interventions: Device: Crosslinked Hyaluronic Acid (CLHA) Hydrogel with and without Lidocaine
- Crosslinked Hyaluronic Acid (CLHA) Hydrogel without Lidocaine (Experimental): Patients were treated, on the other side of the face with crosslinked Hyaluronic Acid Hydrogel without lidocaine hydrochloride.
  Interventions: Device: Crosslinked Hyaluronic Acid (CLHA) Hydrogel with and without Lidocaine

INTERVENTIONS:
Device: Crosslinked Hyaluronic Acid (CLHA) Hydrogel with and without Lidocaine — The injection should be performed at variable depth of the skin (dermal or subdermal), depending on the area to be treated and on the product variants, in accordance to the IFU of the IPs

SUMMARY:
The aim of this interventional, pre-market, double- blinded, controlled, two stages study is to evaluate the performance and safety of Crosslinked Hyaluronic Acid (CLHA) Hydrogel (with and without Lidocaine) for the Treatment of Soft Tissue Deficits.

DETAILED DESCRIPTION:
The performance of Crosslinked Hyaluronic Acid Hydrogel (with and without Lidocaine), for the correction of congenital and acquired deficits of soft tissue, will be evaluated using the change from baseline to V3 in the Wrinkle Severity Rating Scale (WSRS) for 26 mg/ml and 18mg/ml CLHA formulations and in the Lip Fullness Scale (LFS) for 20 mg/ml CLHA formulation.

The duration of the aesthetic effect of Crosslinked Hyaluronic Acid Hydrogel (with and without Lidocaine) for the correction of NLFs, perioral wrinkles and lips augmentation, will be assessed using the mean of the absolute change from baseline to each follow up visit in WSRS and LFS score. WSRS and LFS will be assessed by the evaluating investigator who will be different by the treating investigator.

The aesthetic appearance of the Crosslinked Hyaluronic Acid Hydrogel (with and without Lidocaine) will be assessed using the Global Aesthetic Improvement Scale (GAIS) at each visit. The GAIS will be completed by both the subjects and the evaluating investigators; The volume of material required to achieve an optimal correction result will be assessed at baseline and at optional touch up; The pain intensity after injection of Crosslinked Hyaluronic Acid Hydrogel (with and without Lidocaine) will be assessed using a Numerical Rating Scale (NRS) 2 hours after the injection; The patient satisfaction and the usability of Crosslinked Hyaluronic Acid Hydrogel (with and without Lidocaine) will be evaluated with a specific questionnaire, completed by the Principal Investigator.

The Safety of Crosslinked Hyaluronic Acid Hydrogel (with and without Lidocaine) will be assessed by facial examination and vital signs over the duration of the study. Adverse events and serious adverse events will be collected at each planned visit into a diary dispensed to patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient Informed consent form (ICF) signed
* Female and male subjects aged 18-65 years and in good general health;
* Subjects with Soft Tissue Deficits of the face requiring midface volume restoration;
* Willingness to follow all study procedures, including attending all site visits, tests, and examinations;
* Agreeing to present at each study visit without makeup;
* Accepting to not change their habits regarding food, physical activity, make-up use, facial cosmetics, and cleansing products;
* Willingness to not undergo other procedures involving permanent and nonpermanent aesthetic correction (e.g. chemical peel, dermabrasion, ablative laser resurfacing), non-invasive skin-tightening, botulinum toxin injections, dermal filler injections, mesotherapy, or fat injections during the study period of 12 months;
* Willing to follow indications to not be exposed to make-up, excessive heat (sun, UV tanning sessions, or laser), and extreme temperatures (intense cold, sauna, hammam, etc.) after the treatment and until the complete absorption of swelling and reddening.

Exclusion Criteria:

* Presence of recurrent facial/labial herpes;
* Presence of tendon, bone, or muscular implants near the area of intervention;
* Subjects previously treated with fillers anywhere in the face or neck;
* Subjects who have undergone invasive face or neck surgery;
* Ongoing cutaneous allergies and history of hyper- or hypo-pigmentation in the mouth area, keloid formation, or hypertrophic scarring;
* Subjects with a known allergy or sensitivity to any component of the investigation products;
* Subjects with a known allergy or sensitivity to any component of the anesthetic cream;
* Subjects with active autoimmune disease and subjects immunocompromised or immunosuppressed;
* Diabetes mellitus or uncontrolled systemic diseases (endocrine, hepatic renal, cardiac, pulmonary, neurological disorder);
* Problems with coagulation or anti-coagulating therapies in progress;
* Subjects with acute inflammatory process or infection, active herpes infection, or history of chronic or recurrent infections;
* Current treatment with substances which act on blood fluidity (eg. Aspirin, NSAIDs, Vitamin E), anti-inflammatory drugs, anti-histaminic, topic and systemic corticosteroids, narcotic, antidepressant, immunosuppressive drugs (with the except of contraceptive or hormonal treatment starting more than 1 year ago), drugs able to influence the test results in the investigator opinion;
* Known drug and/or alcohol abuse;
* Mental incapacity that precludes adequate understanding or cooperation;
* Any previous permanent and nonpermanent cutaneous treatment for aesthetic correction e.g. chemical peel, dermabrasion, ablative laser resurfacing, non-invasive skin-tightening, botulinum toxin injections, mesotherapy, or fat injections within 6 months prior to study inclusion;
* Pregnancy or breastfeeding;
* COVID-19 vaccination within one month prior to study inclusion;
* Participation in another investigational study within 1 month prior to study inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-04-02 (Actual); Primary Completion 2023-12-02 (Estimated); Study Completion 2023-12-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the CLHA performance in the nasolabial folds | 6 months
  The performance of Crosslinked Hyaluronic Acid Hydrogel (with and without Lidocaine), for the correction of congenital and acquired deficits of soft tissue in the Nasolabial folds, will be evaluated using the change from baseline to V3 in the Wrinkle Severity Rating Scale (WSRS) for 26 mg/ml CLHA formulation. WSRS is a validated 5-point scale (1 = Absent, 5 = Extreme)
Evaluation of the CLHA performance in the perioral lines | 6 months
  The performance of Crosslinked Hyaluronic Acid Hydrogel (with and without Lidocaine), for the correction of congenital and acquired deficits of soft tissue in the perioral lines, will be evaluated using the change from baseline to V3 in the Wrinkle Severity Rating Scale (WSRS) for 18mg/ml CLHA formulations. WSRS is a validated 5-point scale (1 = Absent, 5 = Extreme)
Evaluation of the CLHA performance in the lips | 6 months
  The performance of Crosslinked Hyaluronic Acid Hydrogel (with and without Lidocaine), for the correction of congenital and acquired deficits of soft tissue in the lips, will be evaluated using the change from baseline to V3 in the Lip Fullness Scale (LFS) for 20 mg/ml CLHA formulation. LFS is a validated 5-point scale (0 = Very Thin, 4 = Full).

SECONDARY OUTCOMES:
Evaluation of the restoring the physiological volumes of the face in the nasolabial folds | 6 months
  The performance of Crosslinked Hyaluronic Acid Hydrogel (with and without Lidocaine) used as intended for restoring the physiological volumes of the face n the nasolabial folds, will be assessed using the change, from baseline to each visit, in the Wrinkle Severity Rating Scale (WSRS) for the 26 mg/ml CLHA formulations. WSRS will be assessed by the evaluating investigator who will be different from the treating investigator. WSRS is a validated 5-point scale (1 = Absent, 5 = Extreme).
Evaluation of the restoring the physiological volumes of the face in the perioral lines | 6 months
  The performance of Crosslinked Hyaluronic Acid Hydrogel (with and without Lidocaine) used as intended for restoring the physiological volumes of the face in the perioral lines, will be assessed using the change, from baseline to each visit, in the Wrinkle Severity Rating Scale (WSRS) for the 18mg/ml CLHA formulations. WSRS will be assessed by the evaluating investigator who will be different from the treating investigator. WSRS is a validated 5-point scale (1 = Absent, 5 = Extreme).
Evaluation of the restoring the physiological volumes of the face in the lips | 6 months
  The performance of Crosslinked Hyaluronic Acid Hydrogel (with and without Lidocaine) used as intended for restoring the physiological volumes of the lips, will be assessed using the change, from baseline to each visit in the Lip Fullness Scale (LFS), for 20 mg/ml CLHA. LFS will be assessed by the evaluating investigator who will be different from the treating investigator. LFS is a validated 5-point scale (0 = Very Thin, 4 = Full).
Evaluation of the duration of the aesthetic effect on the nasolabial folds | 6 months
  The duration of the aesthetic effect of Crosslinked Hyaluronic Acid Hydrogel (with and without Lidocaine) for the correction of NLFs will be assessed using the mean of the absolute change from baseline to each follow up visit in WSRS score. WSRS awill be assessed by the evaluating investigator who will be different by the treating investigator. WSRS is a validated 5-point scale (1 = Absent, 5 = Extreme).
Evaluation of the duration of the aesthetic effect on the perioral lines | 6 months
  The duration of the aesthetic effect of Crosslinked Hyaluronic Acid Hydrogel (with and without Lidocaine) for the correction of perioral lines, will be assessed using the mean of the absolute change from baseline to each follow up visit in WSRS score. WSRS will be assessed by the evaluating investigator who will be different by the treating investigator. WSRS is a validated 5-point scale (1 = Absent, 5 = Extreme).
Evaluation of the duration of the aesthetic effect on the lips | 6 months
  The duration of the aesthetic effect of Crosslinked Hyaluronic Acid Hydrogel (with and without Lidocaine) for the correction of lips augmentation, will be assessed using the mean of the absolute change from baseline to each follow up visit in LFS score. LFS will be assessed by the evaluating investigator who will be different by the treating investigator. LFS is a validated 5-point scale (0 = Very Thin, 4 = Full).
Evaluation of the Global Aesthetic Improvement | 6 months
  To evaluate the performance of Crosslinked Hyaluronic Acid Hydrogel (with and without Lidocaine) to improve aesthetic appearance, the Global Aesthetic Improvement Scale (GAIS) will be assessed at each visit. The GAIS will be completed by both the subjects and the evaluating investigators. The GAIS is a validated 5-point scale (1 = extremely improved, 5 worse).

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Persichetti, Prof., Principal Investigator — Fondazione Policlinico Universitario Campus Bio-Medico Roma
Locations (1):
- Fondazione Policlinico Universitario Campus Bio-medico, Roma, Italy

IPD SHARING:
Plan to Share IPD: No